CLINICAL TRIAL: NCT02536664
Title: RIM - Rituximab in Maintenance
Brief Title: Non-Interventional Study to Examine Rituximab Treatment in Follicular Lymphoma Participants
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22283
Record Dates: First submitted 2015-08-24; First posted 2015-09-01 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- First-line Stratum: Participants who were untreated and decided by the treating physician to be treated with Rituximab for the CD 20-positive follicular lymphoma condition.
  Interventions: Drug: Rituximab
- Relapsed/Refractory Stratum: Participants who relapsed after treatment with chemotherapeutic regimens with or without Rituximab and were decided by the treating physician to be treated with Rituximab for the CD 20-positive follicular lymphoma condition.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab
  Other Names: MabThera®

SUMMARY:
It is a non-interventional study with a duration of approximately 24 months per participant to investigate the therapeutic efficiency, safety and treatment regimens of Rituximab maintenance therapy in daily routine in participants with previously untreated, relapsed or refractory cluster of differentiation 20 (CD20)-positive follicular lymphoma (FL) in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Previously untreated, relapsed or refractory CD 20-positive FL
* Responding to rituximab containing induction therapy (complete response [CR] or partial response [PR])
* To receive rituximab maintenance therapy (decision taken by doctor prior to and independent of this non-interventional study)
* No ineligibility for rituximab

Exclusion Criteria:

Not Applicable (NA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with follicular lymphoma who are to be treated with Rituximab in the maintenance dosing period as decided by the physician
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2009-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Essen, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifteen out of 505 participants were screen failure and excluded from the baseline and safety data sets. Safety Set Overall (SSO) included 490 participants who received at least 1 dose of study drug in/during the maintenance period. Therapy line was not reported for 1 participant and participant flow was reported for 489 participants.
Groups:
- First-line Stratum: Participants who were untreated and decided by the treating physician to be treated with Rituximab for the cluster of differentiation (CD) 20-positive follicular lymphoma condition, were observed for a maximum of 2 years.
- Relapsed/Refractory Stratum: Participants who relapsed after treatment with chemotherapeutic regimens with or without Rituximab and were decided by the treating physician to be treated with Rituximab for the CD 20-positive follicular lymphoma condition, were observed for a maximum of 2 years.
Period: Overall Study
Arm/Group | First-line Stratum | Relapsed/Refractory Stratum
Started | 312 | 177
Completed | 205 | 97
Not Completed | 107 | 80
Not completed — Inadequate completion of documentation | 2 | 4
Not completed — Progression | 13 | 18
Not completed — Death due to lymphoma | 2 | 1
Not completed — Death due to other reason | 3 | 2
Not completed — Intolerability | 8 | 6
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Other | 18 | 24
Not completed — Missing | 53 | 20

BASELINE CHARACTERISTICS:
Population: Reduced Safety Set Overall (rSSO): Included participants who received at least 1 dose of study drug during the maintenance therapy with adequate completion of documentation (primary data lock).
Groups:
- First-line Stratum: Participants who were untreated and decided by the treating physician to be treated with Rituximab for the CD 20-positive follicular lymphoma condition, were observed for a maximum of 2 years.
- Total: Total of all reporting groups
Arm/Group | First-line Stratum | Relapsed/Refractory Stratum | Total
Number analyzed (Participants) | 310 | 173 | 483
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (11.6) | 64.0 (11.0) | 63.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 94 | 265
  Male | 139 | 79 | 218

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Alive and Free From Progressive Disease
Description: Progressive Disease is defined as at least a 20 percent (%) increase in the sum of the longest diameter of target lesions, taking) as reference the smallest sum longest diameter recorded since the treatment started or the appearance of 1 or more new lesions (target and non-target lesions) or the unequivocal progression of existing non-target lesions.
Time Frame: 2 years
Population: Included participants who were considered for the efficacy analysis after 2 years of Rituximab maintenance therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First-line Stratum | Relapsed/Refractory Stratum
Number analyzed (Participants) | 305 | 172
percentage of participants | 88.28 [83.97 to 92.59] | 76.03 [68.79 to 83.28]

2. Secondary Outcome: Median Progression Free Survival (PFS) Time
Description: PFS was defined as the time from the date of the first cycle to the first occurrence of progression of tumor or death from any reason (whichever occurred first). If progression or death was not observed during the study, progression-free survival time was censored by the last documented tumor assessment during the maintenance therapy (latest at the end of study after two years). Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of 1 or more new lesions (target and non-target lesions) or the unequivocal progression of existing non-target lesions. PFS was assessed using Kaplan-Meier estimate.
Time Frame: 2 years
Population: Included participants who were considered for the efficacy analysis after 2 years of Rituximab maintenance therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | First-line Stratum | Relapsed/Refractory Stratum
Number analyzed (Participants) | 305 | 172
months | NA [NA to NA] — The median PFS time and 95% Confidence Interval (CI) could not be estimated due to low number of events (disease progression or death) | NA [NA to NA] — The median PFS time and 95% Confidence Interval (CI) could not be estimated due to low number of events (disease progression or death)

3. Secondary Outcome: Percentage of Participants Who Were Alive
Description: Death for any reason was regarded as an event. Percentage of participants who were alive after 2 years of maintenance therapy with Rituximab was reported.
Time Frame: 2 years
Population: Included participants who were considered for the efficacy analysis after 2 years of Rituximab maintenance therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First-line Stratum | Relapsed/Refractory Stratum
Number analyzed (Participants) | 305 | 172
percentage of participants | 96.89 [94.69 to 99.09] | 95.44 [91.81 to 99.07]

4. Secondary Outcome: Median Overall Survival (OS) Time
Description: Survival was the interval of time from date of first dose of study medication to date of death at any time. Participants who had not died were censored at the date of last contact when they were known to be alive. OS was assessed using Kaplan-Meier estimate.
Time Frame: 2 years
Population: Included participants who were considered for the efficacy analysis after 2 years of Rituximab maintenance therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | First-line Stratum | Relapsed/Refractory Stratum
Number analyzed (Participants) | 305 | 172
months | NA [NA to NA] — The median OS and 95% confidence interval (CI) were not estimated due to low number of deaths during the study | NA [NA to NA] — The median OS and 95% CI were not estimated due to low number of deaths during the study

5. Secondary Outcome: Percentage of Participants With Response (Complete Response [CR], Partial Response [PR], Stable Disease [SD] or Progressive Disease [PD] at the End of Maintenance Therapy
Description: CR is defined as the disappearance of all target and non-target lesions and normalization of tumor marker level; PR is defined as at least a 30 percentage (%) decrease in the sum of the longest diameter of target lesions, taking as reference the screening sum longest diameter; SD for target lesions is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started and SD for non-target lesions defined as persistence of 1 or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits. PD is defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of 1 or more new lesions (target and non-target lesions) or the unequivocal progression of existing non-target lesions.
Time Frame: 2 years
Population: Included participants who were considered for the efficacy analysis after 2 years of Rituximab maintenance therapy.
Measure: Number; unit: percentage of participants
Arm/Group | First-line Stratum | Relapsed/Refractory Stratum
Number analyzed (Participants) | 305 | 172
percentage of participants
  CR | 58.4 | 51.2
  PR | 21.0 | 20.9
  SD | 12.1 | 9.3
  PD | 8.5 | 18.6

6. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: The percentage of participants was presented with respect to the best overall response (CR, PR, SD). CR is defined as the disappearance of all target and non-target lesions and normalization of tumor marker level; PR is defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the screening sum longest diameter; SD for target lesions is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started and SD for non-target lesions defined as persistence of 1 or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: 2 years
Population: Included participants who were considered for the efficacy analysis after 2 years of Rituximab maintenance therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First-line Stratum | Relapsed/Refractory Stratum
Number analyzed (Participants) | 305 | 172
percentage of participants | 98.4 [96.9 to 99.8] | 96.5 [93.8 to 99.3]

7. Secondary Outcome: Percentage of Participants With Initiation of New Therapy
Description: Percentage of participants for whom new therapy was initiated at the end of maintenance therapy was reported.
Time Frame: 2 years
Population: Included participants who were considered for the efficacy analysis after 2 years of Rituximab maintenance therapy.
Measure: Number; unit: percentage of participants
Arm/Group | First-line Stratum | Relapsed/Refractory Stratum
Number analyzed (Participants) | 305 | 172
percentage of participants
  No data | 16.7 | 11.6
  No | 75.7 | 69.2
  Yes | 7.5 | 19.2

ADVERSE EVENTS:
Time Frame: 2 years
Description: SSO, 1 participant was excluded as no therapy line was reported and serious adverse events data was reported for 489 participants. rSSO was used for reporting non-serious adverse events.
Arm/Group | First-line Stratum | Relapsed/Refractory Stratum
Serious Adverse Events (participants affected / at risk) | 35/312 | 39/177
Other Adverse Events (participants affected / at risk) | 0/310 | 30/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | First-line Stratum (N=312) | Relapsed/Refractory Stratum (N=177)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 5 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 5
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Colitis microscopic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Death (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 1 | 0
Pain (General disorders) | 1 | 5
Pyrexia (General disorders) | 3 | 2
Fatigue (General disorders) | 0 | 1
Ill-defined disorder (General disorders) | 0 | 1
Performance status disorder (General disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Immunodeficiency (Immune system disorders) | 0 | 1
Bacterial infection (Infections and infestations) | 2 | 4
Bronchiolitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Haemophilus sepsis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 3 | 7
Viral infection (Infections and infestations) | 2 | 1
Anal abscess (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Infectious colitis (Infections and infestations) | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
B-lymphocyte count decreased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Blast cells present (Investigations) | 0 | 1
Carbohydrate antigen 15-3 increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | First-line Stratum (N=310) | Relapsed/Refractory Stratum (N=173)
Leukopenia (Blood and lymphatic system disorders) | 0 | 21
Bacterial Infection (Infections and infestations) | 0 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.